PRINCIPAL INVESTIGATOR: Mark Roschewski, M.D.

**STUDY TITLE:** Phase 1 Study of Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, and Revlimid (VIPOR) for Diffuse Large B-cell lymphoma involving the Central Nervous System

STUDY SITE: NIH Clinical Center

Cohort: Screening - Affected Patient

Consent Version: 09/01/2022

## WHO DO YOU CONTACT ABOUT THIS STUDY?

Mark Roschewski, M.D.

## KEY INFORMATION ABOUT THIS RESEARCH

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). This section provides the information we believe is most helpful and important to you in making your decision about participating in this study. Additional information that may help you decide can be found in other sections of the document. Taking part in research at the NIH is your choice.

You are being asked to take part in this study because you have B-cell lymphoma in central nervous system (CNS) that does not respond to treatment or response to treatment does not last very long or there is no standard treatment for you.

The main purpose of this research study is to learn if it is safe to give individuals with these cancers the drugs: venetoclax, ibrutinib, prednisone, obinutuzumab, and lenalidomide (VIPOR). We also hope to learn if this combination of drugs may work in the treatment of aggressive B-cell lymphomas with involvement of the central nervous system (CNS).

The drugs in the VIPOR regimen have each been approved and used either alone or in combination to treat types of lymphoma, however the use and combination of the drugs in this study is investigational. An "investigational drug" is a drug or combination of drugs that is being tested and is not approved in the United States by the U.S. Food and Drug Administration (FDA).

There are other drugs and treatments, such as other chemotherapy regimens, radiation therapy, single-agent targeted therapy and/or approved forms of immunotherapy, that may be used for treatment of your disease. These can be prescribed by your regular cancer doctor if you are not in this study. These drugs all work in different ways in the body as compared to the study drugs and with different side effects. If you would prefer other drugs or treatments, you should consider not joining this study.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 09/01/2022


IRB NUMBER: 000516

IRB APPROVAL DATE: 11/09/2022

This consent is for "screening." We would like to find out if you are able to take part in this study.

This will involve evaluation of your health history, physical exam, having standard blood tests, scans, and test of your heart. You also may have lumbar puncture and biopsy of your tumor if we need them for confirmation of your diagnosis.

Screening involves only standard clinical tests, so we do not think you may experience serious side effects during screening.

There may be no direct benefit to you from taking part in the study. However, you may gain clinical information about your disease, or your organ function that will be helpful to your overall medical care. If you would like, we can share the results of these screening tests and notes with your personal physician.

The screening portion of this study will take about a week. You can stop screening at any time.

The remaining document will now describe the research study in more detail. This information should be considered before you make your choice. Members of the study team will talk with you about the information in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research interventions in which they would want to participate. Take the time you need to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

If the individual being asked to participate in this research study is not able to give consent for themselves, you, as the Legally Authorized Representative, will be their decision-maker and you are being asked to give permission for this person to be in this study. For the remainder of this document, the term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

## WHY IS THIS STUDY BEING DONE?

This part of the study is to determine if you are suited for the treatment part of this study.

You are being asked to take part in this study because you have B-cell lymphoma in central nervous system (CNS) which may be treated with the combination of drugs on the treatment study.

#### WHAT WILL HAPPEN DURING THE STUDY?

All of these tests or procedures are part of your regular care. If you have had some of these tests or procedures recently, they may or may not have to be repeated. The following tests and procedures are needed to determine whether you are eligible for this trial:

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


- Medical history: A complete review of your medical history, including obtaining
  information about your diagnosis and previous treatments, and reviewing information
  about your other conditions. If you have medical records from another clinic or hospital,
  you will be asked to get copies of these records, or your study doctor may be able to request
  them on your behalf.
- Physical exam: This will include taking your weight, vital signs (temperature, blood pressure, heart rate, breathing rate), seeing how you function in your daily activities, any current symptoms of your condition and a review of all medications that you take
- Standard blood and urine tests:
  - Tests to measure your liver, kidney, white blood cells, red blood cells and platelets, blood electrolytes and how well your blood clots
  - If you are a woman able to get pregnant and you are not already known to be pregnant, you will also have a pregnancy test done. This may be done by blood or urine test. You will not be able to participate if you are pregnant.
  - To check for Hepatitis B and C infection
  - To check for HIV infection: As part of this study, we will test you for infection with the human immunodeficiency virus (HIV), the virus that causes AIDS. If you are infected with HIV you will not be able to participate in this study. We will tell you what the results mean, how to find care, how to avoid infecting others, how we report HIV infection, and the importance of informing your partners at possible risk because of your HIV infection
- Imaging to show all sites of disease, including
  - Computer tomography (CT) scan, a series of x-ray images of your chest, abdomen and pelvis,
  - ➤ 18F FDG PET scan. A Positron Emission Tomography scan or PET scan for short lets doctors see the activity of cells in specific tissues of the whole body. A sugar, which is attached to a chemical that gives off a signal, is injected into you intravenously before the scan. The scanner records the signals through the body.
  - ➤ MRI (magnetic resonance imaging): MRI uses a strong magnetic field and radio waves to take pictures of the body. We will obtain pictures of your brain for this study. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, you will lie on a table that can slide in and out of the cylinder. We will place soft padding or a coil around your head. You will be in the scanner about 45 minutes. You may be asked to lie still for up to 15 minutes at a time. While in the scanner you will hear loud knocking noises, and you will be fitted with earplugs or earmuffs to muffle the sound. You will be able to communicate with the MRI staff at all times during your scan, and you may ask to be moved out of the machine at any time.

It is very important that you do not move your head or body inside the scanner. We will use padding around your head to help keep it in place.

We may place a bar in your mouth to help keep your head still.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


- An electrocardiogram (EKG) of the heart will be done to check the electrical activity and the function of your heart.
- Lumbar puncture ("spinal tap") or Ommaya tap to take cerebral spinal fluid (CSF) samples. Lumbar puncture involves inserting a small needle into your lower back to sample CSF. If you have an Ommaya reservoir, an Ommaya tap is when a small needle is inserted into the small reservoir under the skin of your scalp to sample CSF.
- A sample of tissue from any previous surgery or biopsy will be tested at NCI to confirm your diagnosis, stage, and status of your disease. If no tissue is available, then a biopsy may need to be performed if you have accessible tumor site. Usually, tissue can be obtained safely and comfortably with local anesthesia. If you require conscious sedation before undergoing a biopsy, you will be informed of the risks and you will be asked to sign an additional consent prior to undergoing the procedure.
- Lenalidomide Revlimid REMS<sup>TM</sup> Program Participation

You have been informed of the risk of birth defects. If you are female, you agree not to become pregnant while taking lenalidomide. For this reason, lenalidomide is provided to patients under a special distribution program called REVLIMID REMS®.

In order to participate in this study, you must register into and follow the requirements of the Revlimid REMS<sup>TM</sup> program of Celgene Corporation. This program provides education and counseling on the risks of lenalidomide, including fetal exposure, blood clots and reduced blood counts. You will be required to receive counseling every 28 days, or more frequently dependent on treatment regimen, during treatment with lenalidomide, follow the pregnancy testing and birth control requirements of the program that are appropriate for you and take telephone surveys regarding your compliance with the program.

By signing this consent, you understand and agree to receive counseling and to comply with the pregnancy precaution requirements of the REVLIMID REMS<sup>TM</sup> program. You will be registered in the REVLIMID REMS<sup>TM</sup> program.

In order to obtain lenalidomide free of charge from Celgene, your name, address, phone, date of birth and the fact that you are participating in this trial will be disclosed to Celgene and its agents or vendors that supply lenalidomide and administer the REVLIMID REMS® program. By signing this consent form, you agree to this disclosure.

The study staff will provide you with more information about this program. It is required of all patients who receive lenalidomide whether on or off a study.

## HOW LONG WILL THE STUDY TAKE?

If you agree to take part in this study, your involvement is expected to require about a week on the screening portion.

#### HOW MANY PEOPLE WILL PARTICIPATE IN THIS STUDY?

We plan to have approximately 16 people participate in this study at the NIH.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


## WHAT ARE THE RISKS AND DISCOMFORTS OF BEING IN THE STUDY?

- Blood draws (about 2.1 tablespoons will be collected at most during a visit): The possible side effects of drawing blood include pain, bleeding, bruising, dizziness, lightheadedness, fainting and, on rare occasions, local blood clot formation or infection with redness and irritation of the vein.
- Urine collection: There are no known physical risks of collecting urine.
- Tumor biopsy (if needed): The likely side effects include discomfort or pain, redness, swelling, and/or bruising at the site of the needle insertion. Bleeding from the site of the needle insertion is a less likely risk. Rarely, significant infection or bleeding from this procedure, allergic reaction to the anesthetic, or formation of a scar at the site of needle entry occurs. If you will have sedation with the procedure, these risks will be discussed with you prior to the procedure. You will be asked to sign a separate consent form prior to any biopsy procedure.
- EKG: Some skin irritation can occur where the EKG (also referred to as ECG) electrodes are placed. Once the electrodes are placed, the test will begin, is completely painless, and generally takes less than a minute to perform. After the test, the electrodes are removed.
- Lumbar puncture: The lumbar puncture (LP) may cause pain at the site where the needle goes in and the spinal fluid is taken. There is a small risk of infection or bleeding. After the lumbar puncture you may get a headache. About a third of adults report a headache after an LP. To minimize the risk of a headache, the doctor will use a small needle and may prescribe bed rest for one or more hours after the procedure. If a headache occurs, it is usually mild and can be controlled by bed rest, drinking lots of fluids and a pain pill, such as acetaminophen. Rarely, the headache is severe and may require additional treatment with a "blood patch". In this procedure, a small amount of your own blood is injected into the lumbar puncture site. This procedure is generally effective in stopping the headache. A rare but serious complication of a LP, if it is done when the pressure inside the head is higher than normal (such as when a brain tumor is present), is known as medullary herniation which can result in death. Increased intracranial pressure is very unlikely to be present. The LP will not be done if there are any clinical indications that you have increased intracranial pressure, a skin infection in the lower back area, or bone malformation of the lower back (including severe scoliosis) which would make a LP difficult. To minimize these risks, the lumbar puncture procedure will be performed by a medical professional specifically trained to do this procedure.
- Fluid Collection by Ommaya Reservoir: Withdrawing spinal fluid from an Ommaya Reservoir conveys a small risk of infection and a minor amount of discomfort from the needle puncture.
- CT and PET scans: If contrast dye is used, there is a risk for allergic reaction to the dye. Participants might experience hives, itching, headache, difficulty breathing, increased heart rate, and swelling. If you are allergic to or sensitive to medications, contrast dye, iodine, or shellfish, please notify your study doctor. If you have had kidney failure or other kidney problems in the past, please notify your study doctor

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


MRI (magnetic resonance imaging): People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have. In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away. There are no known long-term risks of MRI scans.

Risk for gadolinium enhanced MRI scans:

**Procedure:** During part of the MRI you may receive gadolinium, a contrast agent, through an intravenous (iv) catheter. It will be done for medical purposes.

**Risks:** The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives, and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis" which has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is not normal or if you received gadolinium within the previous month.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA recently issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


Some types of gadolinium contrast drugs are less likely to remain than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain.

We will also give you additional information called a "Medication Guide." Upon request, we will give you individual information about retained gadolinium we see on your studies.

## What are the risks of radiation from being in the study?

During your participation in the screening portion of this study, you will be exposed to radiation from one CT scan of the chest, abdomen and pelvis and one 18F-FDG PET scan. The amount of radiation exposure you will receive from these procedures is equal to approximately 2.3 rem. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

The CT and PET scans that you get in this study will expose you to roughly the same amount of radiation as 7.7 years' worth of background radiation. Most of the time, this amount of extra radiation is not harmful to you. However, scientists believe that being exposed to too much radiation can cause harmful side effects. This could include getting a new cancer. We estimate that this could happen in about 1 out of every 1000 people who get a very large amount of extra radiation.

You may not participate in this study if you are pregnant. If you are able to become pregnant, we will perform a pregnancy test before exposing you to radiation. You must tell us if you may have become pregnant within the previous 14 days because the pregnancy test is unreliable during that time.

## WHAT ARE THE BENEFITS OF BEING IN THE STUDY?

You might not benefit from being in this study.

However, you may gain clinical information about your disease or your organ function that will be helpful to your overall medical care. This testing may make you eligible to participate in this research study at the NIH If you would like, the results of these screening tests and procedures will be communicated to your personal physician.

## Are there any potential benefits to others that might result from the study?

In the future, other people might benefit from this study because of the knowledge that will be gained.

## WHAT OTHER OPTIONS ARE THERE FOR YOU?

Before you decide whether or not to be in this study, we will discuss other options that are available to you. Instead of being in this study, you may choose not to be screened.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


## **DISCUSSION OF FINDINGS**

## New information about the study

If we find out any new information that may affect your choice to participate in this study, we will get in touch with you to explain what we have learned. This may be information we have learned while doing this study here at the NIH or information we have learned from other scientists doing similar research in other places.

#### Return of research results

The results of the standard tests performed as part of the research are available to you as part of your medical record.

## EARLY WITHDRAWAL FROM THE STUDY

You will be removed from the study if:

• You are found not to be eligible for the study

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases cannot be recalled and destroyed.

# STORAGE, SHARING AND FUTURE RESEARCH USING YOUR SPECIMENS AND DATA

## Will your specimens or data be saved for use in other research studies?

As part of this study, we are obtaining specimens and data from you. We will remove all the identifiers, such as your name, date of birth, address, or medical record number and label your specimens and data with a code so that you cannot easily be identified. However, the code will be linked through a key to information that can identify you. We plan to store and use these specimens and data for studies other than the ones described in this consent form that are going on right now, as well as studies that may be conducted in the future. These studies may provide additional information that will be helpful in understanding B-cell lymphoma or other diseases or conditions. This could include studies to develop other research tests, treatments, drugs, or devices, that may lead to the development of a commercial product by the NIH and/or its research or commercial partners. There are no plans to provide financial compensation to you if this happens. Also, it is unlikely that we will learn anything from these studies that may directly benefit you.

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


| I give permiss described abo | sion for my coded specimens and data to be stored and used for future research as eve. |
|---|---|
| Yes | No |
| Initials | |
| Will your spe | ecimens or data be shared for use in other research studies? |
| maintain the o | e your coded specimens and data with other researchers. If we do, while we will code key, we will not share it, so the other researchers will not be able to identify hay be doing research in areas that are similar to this study or in other unrelated researchers may be at NIH, other research centers and institutions, or commercial |
| | sion for my coded specimens and data to be shared with other researchers and used archers for future research as described above. |
| Yes Initials | No |
| initiais | initials |

If you change your mind and do not want us to store and use your specimens and data for future research, you should contact the research team member identified at the top of this document. We will do our best to comply with your request but cannot guarantee that we will always be able to destroy your specimens and data. For example, if some research with your specimens and data has already been completed, the information from that research may still be used. Also, for example, if the specimens and data have been shared already with other researchers, it might not be possible to withdraw them.

In addition to the planned use and sharing described above, we might remove all identifiers and codes from your specimens and data and use or share them with other researchers for future research at the NIH or other places. When we or the other researchers access your anonymized data, there will be no way to link the specimens or data back to you. We will not contact you to ask your permission or otherwise inform you before we do this. We might do this even if you answered "no" to the above questions. If we do this, we would not be able to remove your specimens or data to prevent their use in future research studies, even if you asked, because we will not be able to tell which are your specimens or data.

NIH policies require that your clinical and other study data be placed in an internal NIH database that is accessible to other NIH researchers for future research. Usually, these researchers will not have access to any of your identifiers, such as your name, date of birth, address, or medical record number; and your data will be labeled with only a code. We cannot offer you a choice of whether your data to be placed in this database or not. If you do not wish to have your data placed in this database, you should not enroll in this study.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


## How long will your specimens and data be stored by the NIH?

Your specimens and data may be stored by the NIH indefinitely.

## Risks of storage and sharing of specimens and data

When we store your specimens and data, we take precautions to protect your information from others that should not have access to it. When we share your specimens and data, we will do everything we can to protect your identity, for example, when appropriate, we remove information that can identify you. Even with the safeguards we put in place, we cannot guarantee that your identity will never become known or someone may gain unauthorized access to your information. New methods may be created in the future that could make it possible to re-identify your specimens and data.

#### **PAYMENT**

## Will you receive any type of payment for taking part in this study?

You will not receive any payment for taking part in this study.

## REIMBURSEMENT

## Will you receive reimbursement or direct payment by NIH as part of your participation?

This study does not offer reimbursement for parents and participants, or payment of, hotel, travel, or meals during the screening process.

#### **COSTS**

## Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

## **CONFLICT OF INTEREST (COI)**

The NIH reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

No NIH investigator involved in this study receives payments or other benefits from any company whose drug, product or device is being tested.

## PATIENT IDENTIFICATION

## **Consent to Participate in a Clinical Research Study**

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


## CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database. Your test results will be identified by a unique code and the list that links the code to your name will be kept separate from your sample and health information. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you.

## Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

## **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


- is required to be disclosed by Federal, State, or local laws, for example, when information
  must be disclosed to meet the legal requirements of the federal Food and Drug
  Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

## **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical information that we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

## POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

## PROBLEMS OR QUESTIONS



## CONSENT DOCUMENT

Please keep a copy of this document in case you want to read it again.

## PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


IRB NUMBER: 000516

IRB APPROVAL DATE: 11/09/2022

| Signature of Research Particip | Print Name of Research | Participant Date |
|---|---|---|
| about this study and have been to make research decisions on b | atative (LAR) for an Adult Unable to Congiven the opportunity to discuss it and to as we half of the adult participant unable to conseable, the information in the above consent we oparticipate in the study. | k questions. I am legally authorient and have the authority to prove |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigate | or Date |
| Witness should sign below if 1. A short form consent | process has been used to enroll a non-En | glish speaking subject or |
| Witness should sign below if 1. A short form consent 2. An oral presentation | | glish speaking subject or |
| Witness should sign below if 1. A short form consent 2. An oral presentation Signature of Witness | process has been used to enroll a non-En<br>of the full consent has been used to enroll | glish speaking subject or<br>a blind or illiterate subject Date |
| Witness should sign below if 1. A short form consent 2. An oral presentation Signature of Witness NIH ADMINISTRATIVE INTERPRETER: An interpreter, or other incession | process has been used to enroll a non-En of the full consent has been used to enroll Print Name of Witness | glish speaking subject or a blind or illiterate subject Date GARDING THE USE OF |
| Witness should sign below if 1. A short form consent 2. An oral presentation Signature of Witness NIH ADMINISTRATIVE INTERPRETER: An interpreter, or other income also serve as the witness. An interpreter, or other income also serve as the witness. | Print Name of Witness SECTION TO BE COMPLETED RE dividual, who speaks English and the particip consent and served as a witness. The investigations of the particip consent but did not serve as a witness. The | glish speaking subject or a blind or illiterate subject Date Date Date pant's preferred language facilitate stigator obtaining consent may pant's preferred language facilitate name or ID code of the person |

File in Section 4: Protocol Consent (1) IRB NUMBER: 000516 Version Date: 09/01/2022 IRB APPROVAL DATE: 11/09/2022
